CLINICAL TRIAL: NCT00076037
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a CTL Multi-Epitope Peptide HIV Vaccine Formulated With RC529-SE, With or Without GM-CSF, in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Safety of and Immune Response to a New HIV Vaccine: HIV CTL MEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 056; 10122 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-01-13; First posted 2004-01-14 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; Granulocyte-Macrophage Colony-Stimulating Factor; AIDS Vaccines; HIV-1; HIV Seronegativity; Injections, Intramuscular; RC529; Epitopes; T-Lymphocytes, Cytotoxic
MeSH Terms: conditions — HIV Infections | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Biological: HIV CTL MEP administered with RC529-SE adjuvant
Drug: GM-CSF

SUMMARY:
The effectiveness of a vaccine can be improved by using a "prime boost strategy" or by using an adjuvant. A prime boost strategy is the administration of one type of vaccine (the primer) followed by the administration of another type vaccine (the booster). An adjuvant is a substance that can enhance the immune response when given at the same time as a vaccine.

This study will evaluate the safety of and immune response to a vaccine designed to be used as part of a prime boost strategy. The study will also evaluate the vaccine when given with an adjuvant. The vaccine in this study is not produced from live HIV or from infected cells. It does not contain HIV, and it cannot cause HIV infection.

DETAILED DESCRIPTION:
Prime-boost vaccine strategies are aimed at inducing different types of immune responses and enhancing the overall immune response, a result that may not occur with a single type of vaccine. This trial will evaluate the safety and immunogenicity of an HIV multi-epitope peptide cytotoxic T lymphocyte (HIV CTL MEP) vaccine developed as part of a prime-boost strategy and designed to be administered in combination with an HIV DNA vaccine.

The HIV CTL MEP vaccine is a mixture of four synthetic peptides, each containing one of three different HIV CTL epitopes derived from env or gag. The use of multiple conserved CTL epitopes will address the extraordinary diversity found among HIV strains. The vaccine is administered with RC529-SE, an analogue of monophosphoryl lipid A. The vaccine/adjuvant combination will be evaluated with or without coadministration of granulocyte-macrophage colony-stimulating factor (GM-CSF).

Participants will be randomly assigned to receive either the vaccine with the RC529-SE adjuvant, the vaccine with both adjuvants (RC529-SE and GM-CSF), or a placebo. The vaccine, adjuvants, and placebo will all be given as an injection into the upper arm. Participants will have 11 study visits. Study visits will include a physical exam, medical interview, and blood and urine tests. Participants will receive an injection at three of these visits: study entry and Months 1 and 3. Participants will be followed for 1 year after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Willing to receive HIV test results
* Good general health
* One of the following major histocompatibility (MHC) alleles: HLA A3, B7, or B8
* Acceptable methods of contraception for females of reproductive potential
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive
* Access to participating site and available for follow-up during the 15 month study

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Serious adverse reaction to a vaccine. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Hypersensitivity to egg products or yeast-derived products
* Autoimmune disease or immunodeficiency
* Active syphilis
* Unstable asthma
* Type 1 or Type 2 diabetes mellitus
* Thyroid disease requiring treatment in the past 12 months
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2004-04; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spearman, MD, Study Chair — Vanderbilt University; Spyros Kalams, MD, Study Chair — Vanderbilt University
Locations (7):
- United States (7):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research,Project SAVE-Baltimore, Baltimore, Maryland
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Somani J, Lonial S, Rosenthal H, Resnick S, Kakhniashvili I, Waller EK. A randomized, placebo-controlled trial of subcutaneous administration of GM-CSF as a vaccine adjuvant: effect on cellular and humoral immune responses. Vaccine. 2002 Dec 13;21(3-4):221-30. doi: 10.1016/s0264-410x(02)00463-2. PMID 12450697
- [Background] Gilbert PB, Chiu YL, Allen M, Lawrence DN, Chapdu C, Israel H, Holman D, Keefer MC, Wolff M, Frey SE; NIAID HIV Vaccine Trials Network. Long-term safety analysis of preventive HIV-1 vaccines evaluated in AIDS vaccine evaluation group NIAID-sponsored Phase I and II clinical trials. Vaccine. 2003 Jun 20;21(21-22):2933-47. doi: 10.1016/s0264-410x(03)00158-0. PMID 12798637